CLINICAL TRIAL: NCT06426628
Title: Clinical Utility of Management of Patients With CT and LDCT Identified Pulmonary Nodules Using the Percepta Nasal Swab Classifier
Brief Title: Clinical Utility of Management of Patients With Pulmonary Nodules Using the Percepta Nasal Swab Classifier
Acronym: NIGHTINGALE
Status: Recruiting | Type: Observational
Sponsor: Veracyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF009-050P
Record Dates: First submitted 2024-05-10; First posted 2024-05-23 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Nodule, Solitary; Lung Cancer
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Arm: Percepta Nasal Swab test result will be returned to the physician investigator.
- Control Arm: Percepta Nasal Swab test result will not be returned to the physician investigator.

SUMMARY:
The goal of this observational study is to learn how a physician uses the results of the Percepta® Nasal Swab test to manage people with a newly identified pulmonary nodule.

The main questions it aims to answer are:

* Does the use of the Percepta Nasal swab test reduce the number of invasive procedures in people with a low-risk result and whose nodule is benign?
* Does the use of the Percepta Nasal swab test decrease the time to treatment in people with a high-risk result and whose nodule is cancer?

Participants will be randomly assigned to either a group where the test result is provided to the physician (test arm) or to a group where the test result is not provided (control arm). Researchers will compare management of participants in the two groups.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized study to evaluate the clinical utility of the Percepta® Nasal Swab classifier in managing patients with pulmonary nodules identified incidentally or by lung cancer screening. Patients will be randomized to either the test group, where the test result will be returned to the physician to incorporate into decision-making on how to manage the patient's nodule, or the control group which will represent the standard of care where the result will not be returned to the physician. The study will observe and evaluate how the addition of the Percepta Nasal Swab classifier result impacts current management of newly identified lung nodules.

The study will enroll approximately 2400 participants meeting eligibility criteria at up to 100 centers in the US. Enrollment is expected to take approximately 24 months and participants will be followed for 24 to 30 months or until a diagnosis of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate nasal epithelial specimen collection
* Signed written Informed Consent obtained
* Subject clinical history available for review by sponsor and regulatory agencies
* New nodule identified on imaging < 90 days prior to nasal sample collection
* CT report available for index nodule
* 29 - 85 years of age
* Current or former smoker (>100 cigarettes in a lifetime)
* Pulmonary nodule ≤30 mm detected by CT

Exclusion Criteria:

* Active cancer (other than non-melanoma skin cancer)
* Prior primary lung cancer (prior non-lung cancer acceptable)
* Prior participation in this study (i.e., subjects may not be enrolled more than once)
* Current active treatment with an investigational device or drug
* Patient enrolled or planned to be enrolled in another clinical trial that may influence management of the patient's nodule
* Concurrent or planned use of tools or tests for assigning lung nodule risk of malignancy other than clinically validated risk calculators

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current or former smokers (>100 cigarettes in a lifetime) who are 29 - 85 years of age with a newly identified pulmonary nodule ≤30 mm detected by CT
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of invasive diagnostic procedures | From date of randomization until the date the nodule is diagnosed as benign or demonstrates up to 24 months radiographic stability or resolution, assessed up to a total of 30 months.
  Invasive diagnostic procedures performed in the diagnostic workup of newly identified nodules that are benign.

SECONDARY OUTCOMES:
Time to treatment | From date of randomization until the date of first documented treatment for lung cancer, assessed up to a total of 30 months.
  Time to treatment in the diagnostic workup of newly identified nodules that are primary lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Phillip G Febbo, MD, Study Chair — Veracyte, Inc.
Locations (23):
- United States (22):
  - Trinity Health Of New England, Hartford, Connecticut
  - The Stamford Health/The Stamford Hospital, Stamford, Connecticut
  - Bay Pines VA HCS, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Bruce W. Carter Miami VA Medical Center, Miami, Florida
  - Orlando VA Healthcare System, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lexington VA Health Care System, Lexington, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Saint Lukes Hospital, Kansas City, Missouri
  - Mercy Hospital, Springfield, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Good Samaritan Cancer Center, West Islip, New York
  - PulmonIx, LLC, Greensboro, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
- VA Caribbean Healthcare, San Juan, Puerto Rico